CLINICAL TRIAL: NCT01088386
Title: Zyprexa® Relprevv™ Patient Care Program
Status: Enrolling by invitation | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 12991; F1D-MC-B041 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: All patients who will be receiving Zyprexa Relprevv must be enrolled into the Zyprexa Relprevv Patient Care Program

SUMMARY:
The goal of the Zyprexa Relprevv Patient Care Program is to mitigate the risk of negative outcomes associated with Zyprexa Relprevv post-injection delirium/sedation syndrome (PDSS).

DETAILED DESCRIPTION:
The goal of the Zyprexa Relprevv Patient Care Program is to mitigate the risk of negative outcomes associated with Zyprexa Relprevv post-injection delirium/sedation syndrome (PDSS) by:

1. Ensuring Zyprexa Relprevv is prescribed only by certified prescribers, dispensed only by certified dispensers, and dispensed for use only in certified healthcare facilities with ready access to emergency response services, and dispensed for use only with documentation of safe use conditions;
2. Informing health care providers and patients about the risks and the need for continuous observation of patients for at least 3 hours in certified healthcare facilities; and
3. Establishing long-term safety and safe use of Zyprexa Relprevv through periodic monitoring for the risk of PDSS events and by enrolling all patients who receive Zyprexa Relprevv in the Zyprexa Relprevv Patient Care Program registry.

ELIGIBILITY:
Inclusion Criteria:

* Any patients receiving Zyprexa Relprevv enrolled in Zyprexa Relprevv Patient Care Program

Exclusion Criteria:

* Any patient not receiving Zyprexa Relprevv

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical practices in the United States
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2010-03-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence per injection and per patient of post-injection delirium/sedation syndrome (PDSS) events | Baseline to end of study

SECONDARY OUTCOMES:
Type of post-injection delirium/sedation syndrome (PDSS) by clinical presentation and outcome | Baseline to end of study
Potential risk factors of post-injection delirium/sedation syndrome (PDSS). | Baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- United BioSource Corporation, Blue Bell, Pennsylvania, United States